CLINICAL TRIAL: NCT03620552
Title: Safety and Diagnostic Performance of 18F-S16 PET/CT in Healthy Volunteers and Patients With Neurodegenerative Dementia
Brief Title: 18F-S16 PET/CT in Healthy Volunteers and Patients With Neurodegenerative Dementia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oriental Neurosurgery Evidence-Based-Study Team (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S16AD2018
Record Dates: First submitted 2018-07-29; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-06

CONDITIONS: Neurodegenerative Dementia
Keywords: 18F-S16; Neurodegenerative Dementia; PET/CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-S16 injection and PET/CT scan (Experimental): The subjects were intravenously injected with 370MBq 18F-S16 and underwent PET/CT scan immediately after the injection.
  Interventions: Drug: 18F-S16

INTERVENTIONS:
Drug: 18F-S16 — A single dose of nearly 370MBq 18F-S16 were intravenously injected into the subjects immediately before the PET/CT scans

SUMMARY:
This is an open-label dynamic whole-body PET/CT (positron emission tomography/computed tomography) study for investigation of radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of 18F-S16 in healthy volunteers and patients with neurodegenerative dementia.

DETAILED DESCRIPTION:
For interests in clinical translation of 18F-S16, an open-label dynamic whole-body PET/CT study was designed to investigate safety and diagnostic performance of 18F-S16 in patients with neurodegenerative dementia. A single dose of nearly 370 MBq 18F-S16 will be intravenously injected into healthy volunteers and patients with neurodegenerative dementia. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature, routine blood and urine tests, serum alanine aminotransferase, albumin, and creatinine, and any adverse events will be collected from the subjects. Adverse events will also be observed in the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Neurodegenerative Dementia
2. Males and females, ≥40 years old
3. They rely on a combination of neurologic examination and neuropsychological assessment with a battery of tests. Clinical diagnosis was established by sophisticated neurologists.

Exclusion Criteria:

1. Females planning to bear a child recently or with childbearing potential
2. Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
3. Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
4. Known severe allergy or hypersensitivity to IV radiographic contrast.
5. Patients not able to enter the bore of the PET/CT scanner.
6. Inability to lie still for the entire imaging time because of cough, pain, etc.
7. Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
8. Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-10-20 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
Semiquantitative assessment of lesions and biodistribution | One year
  The semiquantitative analysis will be performed by the same physician for all the cases, and the standardized uptake values (SUVs) of brain and other organs will be measured.

SECONDARY OUTCOMES:
Blood pressure | 24 hours
  Systolic and diastolic pressure of subjects will be measured at three time points: right before injection, after scanning, and 24 hours after treatment.
Pulse | 24 hours
  Pulse will be measured at three time points for each subjects: right before injection, after scanning, and 24 hours after treatment.
Respiration frequency | 24 hours
  Respiration frequency will be measured at three time points for subjects: right before injection, after scanning, and 24 hours after treatment.
Temperature | 24 hours
  Temperature will be measured at three time points for subjects: right before injection, after scanning, and 24 hours after treatment.
Serum alanine aminotransferase | 24 hours
  Serum alanine aminotransferase of subjects will be measured at two time points: right before injection and 24 hours after treatment.
Serum albumin | 24 hours
  Serum albumin of subjects will be measured at two time points: right before injection and 24 hours after treatment.
Serum creatinine | 24 hours
  Serum creatinine of subjects will be measured at two time points: right before injection and 24 hours after treatment.
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of subjects will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Li Cai, MD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- PET/CT center,Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China